CLINICAL TRIAL: NCT00456430
Title: Serotonin Transporter Genetic Variation and Amygdalar Activation Correlates of Antidepressant Response
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Responsible Party: Amit Anand, M.D., Indiana University School of Medicine Department of Psychiatry
Organization: Indiana University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0408-34; 41-869-41
Record Dates: First submitted 2005-09-14; First posted 2007-04-05 (Estimated); Last update posted 2011-11-15 (Estimated); Status verified 2010-01

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Escitalopram — 10 mg a day of escitalopram by mouth per day for 4 weeks. Dose may be increased to 20 mg a day after the 4th week depending on tolerance and treatment response.
  Other Names: lexapro

SUMMARY:
The purpose of this study is to find out what parts of the brain have increased or decreased activity when people are depressed and how antidepressant medicine changes this activity in depressed patients.In particular, this study will investigate whether variation in the serotonin transporter gene can affect the response to escitalopram as measured by clinical interview and MRI scan. We will measure activity in different parts of the brain, while subjects see pictures, using Magnetic Resonance Imaging (MRI) scan. There will be three MRI scans; one before we start any medication, one during the study after 3 weeks of treatment and one after six more weeks of treatment. Treatment will consist of Escitalopram. Additionally a blood sample will be taken for genetic testing. The genetic samples collected are to look at variation in a gene (serotonin transporter gene), which affects the functioning of the chemical serotonin in the brain.

DETAILED DESCRIPTION:
Hypotheses:

Hypothesis 1: Depressed patients with the s/s or s/L alleles of the 5-HTTLPR polymorphism will have greater amygdalar activation and decreased cortico-amygdala connectivity compared to patients with L/L genotype

Hypothesis 2: After 2 and 8 weeks of treatment with escitalopram (10 mg) depressed patients with the L/L allele will have a greater decrease in amygdalar activation and a greater increase in cortico-amygdala connectivity than patients with s/s or s/L genotypes.

Methods:

We will stratify the subjects in the two genotype groups so that they are comparable in terms of age and gender distributions. Only depressed patients will be treated with escitalopram. Healthy subjects and unmedicated currently euthymic depressed patients will have baseline scan and subsequent repeat fMRI scans at the same intervals as the depressed patients but will not receive any treatment. After completing the first fMRI scan, depressed patients will undergto one week of single blind placebo lead in. After the first week patient's depression symptoms will be assessed again. If depression symptoms are much better after the first week ( > 20% reduction in HAM-D scores) then the patient will not be asked to do the rest of the study and will be referred to a clinician of their choice for further treatment as necessary. If their depression symptoms do not show much improvement after the first week then they will be asked to take escitalopram for the next 8 weeks. At the end of 3 weeks of treatment from baseline, the patient will undergo a second fMRI scan. Following the second fMRI scan the patient will be continued on escitalopram for another 6 weeks.

ELIGIBILITY:
Inclusion Criteria:Inclusion criteria for Depressed Subjects

1. Ages 18-45 years and able to give voluntary informed consent.
2. Satisfy criteria for Major Depression using the Structured Clinical Interview for DSM-IV (SCID-IV).
3. 17-item Hamilton Depression Rating Scale score > 18
4. Satisfy criteria to undergo an MRI scan based on MRI screening questionnaire
5. Able to be managed as outpatients for initial assessment and during treatment as ascertained by the following -
6. Symptoms not worsening by more than 5 point on either the HDRS during the course of the study.
7. No danger to self or others.
8. No psychotic symptoms.
9. If genetically the patient is a match/meets our requirements for the study. The ratio of s genotype and the l/l genotype is 3:2. Therefore, at some stage in the study we may have more of one type of genotype and may not be able to include a patient for whose genotype we already have sufficient number of subjects.

Inclusion criteria for healthy subjects:

1. Ages 18-60 years and able to give voluntary informed consent.
2. No history of psychiatric illness or substance abuse or dependence as assessed by SCID for non-patients (SCID-NP).
3. No significant family history of psychiatric or neurological illness.
4. Not currently taking any prescription or centrally acting medications.
5. No serious medical or neurological illness as assessed by history, physical examination and laboratory examination including CBC and blood chemistry.
6. If genetically the subject is a match/meets our requirements for the study. The ratio of s genotype and the l/l genotype is 4:1. Therefore, at some stage in the study we may have more of one type of genotype and may not be able to include a patient for whose genotype we already have sufficient number of subjects.

Exclusion Criteria:

* Exclusion criteria for patients

  1. Meeting DSM-IV criteria for schizophrenia, schizophreniform disorder, schizoaffective disorder, atypical psychosis, mental retardation, or organic mental (including organic mood) disorder.
  2. Use of neuroleptic past 2 weeks
  3. Use of antidepressants in the past 2 weeks. If on fluoxetine in the past then should not have been on this medication for 4 weeks.
  4. Use of mood stabilizers in the past 2 weeks
  5. Use of benzodiazepines in the past 2 weeks.
  6. Acutely suicidal or homicidal or requiring inpatient treatment.
  7. Meeting DSM-IV criteria for other substance dependence within the past year, except caffeine or nicotine. The criteria will be evaluated by interview and urinary toxicology screening initially and on test days.
  8. Use of alcohol in the past 1 week.
  9. No serious medical or neurological illness as assessed by physical examination and laboratory examination including CBC and blood chemistry.
  10. Current pregnancy or breast feeding.
  11. Metallic implants.
  12. Previously known positive HIV blood test as reported by the subject.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2003-07; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Decrease in amygdalar activation and increase in cortico-amygdala connectivity as shown by fMRI given at baseline and three weeks from baseline and nine weeks from baseline | Started: July 2003 ended August 2007
Improvement in scores on Hamilton Depression Rating Scale | Started July 2003 Ended August 2007

SECONDARY OUTCOMES:
Improvement in scores on the Hamilton Anxiety Rating Scale | Started July 2003 ended August 2007

CONTACTS AND LOCATIONS:
Overall Officials: Amit Anand, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University Adult Psychiatry Clinic, Indianapolis, Indiana, United States